CLINICAL TRIAL: NCT05444101
Title: Optimizing Psychological Treatment for Pain After Breast Cancer: A Factorial Design Study
Brief Title: Optimizing Psychological Treatment for Pain After Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Danish Council for Independent Research (Other)
Responsible Party: Principal Investigator, Bobby Zachariae, Professor, University of Aarhus
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MOST Pain
Record Dates: First submitted 2022-06-27; First posted 2022-07-05 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Pain, Chronic; Breast Cancer
Keywords: Breast Cancer; Pain; Contemporary cognitive behavioral therapy; Mindful attention; Decentering; Values and committed action; The Multiphase Optimization Strategy (MOST); Psychological pain treatment; Treatment mediators
MeSH Terms: conditions — Chronic Pain; Breast Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: The study uses a 2^3 factorial design, randomizing participants to 8 experimental conditions. The seven active conditions consist of one, two, or three different treatment components. Participants receiving two or three treatment components will be randomized to receive them in different order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Waitlist control (No Intervention): Participants randomized to condition 1 are not offered any treatment components immediately upon enrollment, but will be offered a treatment component of own choice at the end of the study. Total number of sessions: 2 (2 contact hours) following study completion.
- Mindful attention (Experimental): Participants randomized to condition 2 will receive the Mindful attention treatment component. Total number of sessions: 2 (2 contact hours).
  Interventions: Behavioral: Mindful attention
- Decentering (Experimental): Participants randomized to condition 3 will receive the Decentering treatment component. Total number of sessions: 2 (2 contact hours).
  Interventions: Behavioral: Decentering
- Values and committed action (Experimental): Participants randomized to condition 4 will receive the Values and committed action treatment component. Total number of sessions: 2 (2 contact hours).
  Interventions: Behavioral: Values and committed action
- Mindful attention + Decentering (Experimental): Participants randomized to condition 5 will receive the Mindful attention treatment component and the Decentering treatment component in different orders. Total number of sessions: 4 (4 contact hours).
  Interventions: Behavioral: Mindful attention; Behavioral: Decentering
- Mindful attention + Values and committed action (Experimental): Participants randomized to condition 6 will receive the Mindful attention treatment component and the Values and committed action treatment component in different orders. Total number of sessions: 4 (4 contact hours).
  Interventions: Behavioral: Mindful attention; Behavioral: Values and committed action
- Decentering + Values and committed action (Experimental): Participants randomized to condition 7 will receive the Decentering treatment component and the Values and committed action treatment component in different orders. Total number of sessions: 4 (4 contact hours).
  Interventions: Behavioral: Decentering; Behavioral: Values and committed action
- Mindful attention + Decentering + Values and committed action (Experimental): Participants randomized to condition 8 will receive the Mindful attention treatment component, the Decentering treatment component, and the Values and committed action treatment component in different orders. Total number of sessions: 6 (6 contact hours).
  Interventions: Behavioral: Mindful attention; Behavioral: Decentering; Behavioral: Values and committed action

INTERVENTIONS:
Behavioral: Mindful attention — The Mindful attention treatment component consists of a breathing exercise and is operationalized as two sessions (1 hour each) delivered over two weeks, i.e., one session per week, with homework between sessions. Sessions will be delivered online.
  Arms: Mindful attention; Mindful attention + Decentering; Mindful attention + Decentering + Values and committed action; Mindful attention + Values and committed action
Behavioral: Decentering — The Decentering treatment component consists of a guided imagery exercise and is operationalized as two sessions (1 hour each) delivered over two weeks, i.e., one session per week, with homework between sessions. Sessions will be delivered online.
  Arms: Decentering; Decentering + Values and committed action; Mindful attention + Decentering; Mindful attention + Decentering + Values and committed action
Behavioral: Values and committed action — The Values and committed action treatment component consists of identification of personal values and committed action, and is operationalized as two sessions (1 hour each) delivered over two weeks, i.e., one session per week, with homework between sessions. Sessions will be delivered online.
  Arms: Decentering + Values and committed action; Mindful attention + Decentering + Values and committed action; Mindful attention + Values and committed action; Values and committed action

SUMMARY:
The present study aims to optimize psychological treatment for pain after breast cancer by identifying active treatment components. Specifically, a factorial design will be used to evaluate the efficacy and change processes of three psychological treatment components, which have been shown to be efficacious in the treatment of pain after breast cancer.

DETAILED DESCRIPTION:
There is a need for optimization of psychological treatment of pain after breast cancer. Optimization relies on knowledge about the active components of existing treatments. Guided by the Multiphase Optimization Strategy (MOST), the present study aims to address this challenge by identifying active contemporary cognitive behavioral therapy components for breast cancer-related pain. Consistent with the Optimization phase of the MOST framework, a full factorial design will be used to evaluate the efficacy and change processes of three selected treatment components.The overall hypothesis is that the three components will target key maintaining psychological factors in pain, thus leading to reductions in the primary outcomes of pain intensity and -interference. The treatment components and their hypothesized mechanisms of action are as follows:

1. Mindful attention practices will increase attentional control (i.e., the ability to intentionally focus and intentionally shift one's attention), thereby reducing pain hypervigilance, leading to reductions in pain intensity and -interference.
2. Decentering practices will reduce fusion with thoughts (i.e., getting caught up in one's thoughts, feelings and inner experiences), thereby reducing pain catastrophizing, leading to reductions in pain intensity and -interference.
3. Values and committed action (i.e., behavior congruent with one's values) will increase acceptance of discomfort and reduce avoidant behavior, leading to reductions in pain intensity and -interference.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary breast cancer stage I-III
* Min. 6 months post primary treatment (i.e., surgery, chemotherapy, and/or radiotherapy). Endocrine treatment, e.g., Letrozol or Tamoxifen, and/or Zoledronic acid and/or Herceptin treatment is allowed during study participation
* Pain corresponding to a pain score of >= 3 on pain intensity and/or pain interference measured by 11-point Numeric Rating Scales (NRSs)
* Sufficient ability to communicate in Danish
* Sufficient ability to participate in an online-delivered intervention

Exclusion Criteria:

* Non-curable breast cancer (stage IV)
* Breast cancer recurrence
* Bilateral breast cancer
* Other current cancer disease
* Other primary pain condition (e.g., fibromyalgia)
* Current severe psychiatric disorder (e.g., psychosis) hindering study participation
* Insufficient ability to communicate in Danish
* Insufficient ability to participate in an online-delivered intervention

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (11-point Numeric Rating Scale, NRS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The NRS is a validated, self-report instrument assessing pain intensity during the last week. Answer format range: 0 (no pain) to 10 (worst possible pain); total score range: 0-10. A higher score yields more pain.
Pain interference (the 7-item subscale of the Brief Pain Inventory, BPI) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The BPI is a validated, self-report instrument assessing clinical pain. The BPI pain interference subscale assesses pain interference during the last week across 7 domains, i.e., general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Answer format range: 0 (no interference) to 10 (maximal interference); total score range: 0-10. A higher score yields more pain.

SECONDARY OUTCOMES:
Pain intensity (11-point Numeric Rating Scale, NRS) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  The NRS is a validated, self-report instrument assessing pain intensity during the last week. Answer format range: 0 (no pain) to 10 (worst possible pain); total score range: 0-10. A higher score yields more pain.
Pain intensity (11-point Numeric Rating Scale, NRS) | Every day for 6 days following the first session (Td) for each treatment component
  Pain intensity during the last 24 hours will be assessed every day for 6 days following the first session (Td) for each treatment component using the NRS. Answer format range: 0 (no pain) to 10 (worst possible pain); total score range: 0-10. A higher score yields more pain.
Pain interference (the 7-item subscale of the Brief Pain Inventory, BPI) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  The BPI is a validated, self-report instrument assessing clinical pain. The BPI pain interference subscale assesses pain interference during the last week across 7 domains, i.e., general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Answer format range: 0 (no interference) to 10 (maximal interference); total score range: 0-10. A higher score yields more pain.
Pain interference (1 aggregated item assessing pain interference during the last 24 hours within the 7 domains measured with the Brief Pain Inventory, BPI, interference subscale) | Every day for 6 days following the first session (Td) for each treatment component
  Pain interference during the last 24 hours will be assessed every day for 6 days following the first session (Td) for each treatment component using 1 aggregated item assessing pain interference across the 7 domains measured with the BPI interference subscale, i.e., general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Answer format range: 0 (no interference) to 10 (maximal interference); total score range: 0-10. A higher score yields more pain..
Pain burden (11-point Numeric Rating Scale, NRS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The NRS is a validated, self-report instrument assessing pain burden during the last week. Answer format range: 0 (no burden) to 10 (maximal burden); total score range: 0-10. A higher score yields more pain burden.
Pain burden (11-point Numeric Rating Scale, NRS) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  The NRS is a validated, self-report instrument assessing pain burden during the last week. Answer format range: 0 (no burden) to 10 (maximal burden); total score range: 0-10. A higher score yields more pain burden.
Pain quality (the 22-item pain descriptors from the McGill Pain Questionnaire, MPQ) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The pain descriptors from the MPQ constitutes a validated, self-report instrument assessing pain quality (i.e., pain type, namely continuous pain, intermittent pain, neuropathic pain, affective pain) during the last week. Answer format range: 0 (no pain) to 10 (worst possible pain); total score range: 0-60 (continuous, neuropathic and intermittent pain), 0-40 (affective pain). Higher scores yield more pain.
Pain quality (the 22-item pain descriptors from the McGill Pain Questionnaire, MPQ) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  The pain descriptors from the MPQ constitutes a validated, self-report instrument assessing pain quality (i.e., pain type, namely continuous pain, intermittent pain, neuropathic pain, affective pain) during the last week. Answer format range: 0 (no pain) to 10 (worst possible pain); total score range: 0-60 (continuous, neuropathic and intermittent pain), 0-40 (affective pain). Higher scores yield more pain.
Pain frequency (1 item) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  Pain frequency will be assessed using a single question. Answer format range: 1 (never) to 5 (all the time); total score range: 1-5. Higher scores yield higher pain frequency.
Pain frequency (1 item) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  Pain frequency will be assessed using a single question. Answer format range: 1 (never) to 5 (all the time); total score range: 1-5. Higher scores yield higher pain frequency.
Pain catastrophizing (the 13-item Pain Catastrophizing Scale, PCS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The PCS is a validated, self-report instrument assessing pain catastrophizing. Answer format range: 0 (not at all) to 4 (all the time); total score range: 0-52. Higher scores yield more pain catastrophizing.
Pain catastrophizing (the 13-item Pain Catastrophizing Scale, PCS) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  The PCS is a validated, self-report instrument assessing pain catastrophizing. Answer format range: 0 (not at all) to 4 (all the time); total score range: 0-52. Higher scores yield more pain catastrophizing.
Psychological distress (the 14-item Hospital Anxiety and Depression Scale, HADS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The HADS is a validated, self-report instrument assessing psychological distress during the last week. Answer format range: 0 (not at all or never) to 3 (most or all of the time); total score range 0-42. Higher scores yield more psychological distress.
Psychological distress (the 14-item Hospital Anxiety and Depression Scale, HADS) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  The HADS is a validated, self-report instrument assessing psychological distress during the last week. Answer format range: 0 (not at all or never) to 3 (most or all of the time); total score range 0-42. Higher scores yield more psychological distress.
Fear of cancer recurrence (the 9-item Fear of Cancer Recurrence Inventory, FCRI) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The FCRI is a validated, self-report instrument assessing fear of cancer recurrence during the last month. Answer format range: 0 (not at all) to 4 (a great deal); total score range 0-36. Higher scores yield more fear of cancer recurrence.
Fear of cancer recurrence (the 9-item Fear of Cancer Recurrence Inventory, FCRI) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  The FCRI is a validated, self-report instrument assessing fear of cancer recurrence during the last month. Answer format range: 0 (not at all) to 4 (a great deal); total score range 0-36. Higher scores yield more fear of cancer recurrence.
Well-being (the 5-item WHO-5 Well-Being Index, WHO-5) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The WHO-5 is a validated, self-report instrument assessing current well-being. Answer format range: 0 (at no time) to 5 (all the time); total score range: 0-100. Higher scores yield more well-being.
Well-being (the 5-item WHO-5 Well-Being Index, WHO-5) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  The WHO-5 is a validated, self-report instrument assessing current well-being. Answer format range: 0 (at no time) to 5 (all the time); total score range: 0-100. Higher scores yield more well-being.

OTHER OUTCOMES:
Moderator: Socio-demographic characteristics | Baseline (T1)
  Socio-demographic characteristics will be assessed using single questions (e.g., marital status, income, work status).
Moderator: Clinical characteristics | Baseline (T1)
  Clinical data will be obtained from the register of the national Danish Breast Cancer Group (DCBG), including disease characteristics (e.g., date of diagnosis; endocrine receptor status; menopausal status) and allocated treatment protocol (e.g., type of primary surgery; radiotherapy (yes/no); endocrine therapy (yes/no); Herceptin treatment (yes/no); Zoledronic acid (yes/no)).
Moderator: Treatment expectancy | Baseline (T1)
  Treatment expectancy will be assessed using a single question regarding the extent to which the participant expects that the intervention to reduce pain and increase overall well-being. Answer format range: 1 (not at all) to 5 (a great deal); total score range: 1-5. Higher scores indicate stronger expectations that the intervention will lead to a positive outcome.
Moderator: Therapeutic alliance (the 12-item Working Alliance Inventory, WAI) Revised Short Form | 1 week after last session (Post-intervention, T2)
  The WAI is a validated, self-report instrument assessing therapeutic alliance. Answer format range: 1 (never) to 7 (all the time); total score range: 12-84. Higher scores yield a stronger therapeutic alliance.
Moderator: Homework | Before each session (Ts), 1 week after last session (Post-intervention, T2), and 12 weeks after post-intervention (T2) (follow-up, T3)
  Homework will be assessed with 4 single items related to i) whether homework has been conducted (yes/no), and the ii) type, iii) frequency (number of days per week), and iv) duration of completed homework (average number of minutes per day).
Mediator: Mindful attention (the 15-item Mindful Attention Awareness Scale, MAAS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The MAAS is a validated, self-report instrument assessing individual differences in the frequency of mindful states over time. Answer format range: 1 (almost always) to 6 (almost never); total score range: 1-6. Higher scores yield higher levels of mindful attention.
Mediator: Mindful attention (the 15-item Mindful Attention Awareness Scale, MAAS) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  The MAAS is a validated, self-report instrument assessing individual differences in the frequency of mindful states over time. Answer format range: 1 (almost always) to 6 (almost never); total score range: 1-6. Higher scores yield higher levels of mindful attention.
Mediator: Mindful attention (2 items from the 15-item Mindful Attention Awareness Scale, MAAS) | Before each session (Ts)
  MAAS items 13 and 7 will be assessed before each session (Ts). Answer format range: 1 (almost always) to 6 (almost never). Higher scores yield higher levels of mindful attention.
Mediator: Mindful attention (1 item from the 15-item Mindful Attention Awareness Scale, MAAS) | Every day for 6 days following the first session for each treatment component (Td)
  MAAS item 7 will be assessed every day for 6 days following the first session (Td) for each treatment component. Answer format range: 1 (almost always) to 6 (almost never). Higher scores yield higher levels of mindful attention.
Mediator: Decentering (the 11-item Experiences Questionnaire, EQ) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The EQ is a validated, self-report instrument assessing decentering. Answer format range: 1 (do not agree at all) to 5 (agree completely); total score range: 11-55. Higher scores yield higher levels of decentering.
Mediator: Decentering (the 11-item Experiences Questionnaire, EQ) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  The EQ is a validated, self-report instrument assessing decentering. Answer format range: 1 (do not agree at all) to 5 (agree completely); total score range: 11-55. Higher scores yield higher levels of decentering.
Mediator: Decentering (2 items from the 11-item Experiences Questionnaire, EQ) | Before each session (Ts)
  EQ items 5 and 7 will be assessed before each session (Ts). Answer format range: 1 (do not agree at all) to 5 (agree completely). Higher scores yield higher levels of decentering.
Mediator: Decentering (1 item from the 11-item Experiences Questionnaire, EQ) | Every day for 6 days following the first session for each treatment component (Td)
  EQ item 5 will be assessed every day for 6 days following the first session (Td) for each treatment component. Answer format range: 1 (do not agree at all) to 5 (agree completely). Higher scores yield higher levels of decentering.
Mediator: Pain acceptance and activity engagement (the 20-item Chronic Pain Acceptance Scale, CPAS) | Baseline (T1) to 1 week after last session (Post-intervention, T2)
  The CPAS is a validated, self-report instrument assessing pain acceptance and activity engagement. Answer format range: 0 (never true) to 6 (always true); subscale score range: 0-54 (pain acceptance subscale), 0-66 (activity engagement subscale). Higher scores yield more acceptance and activity engagement.
Mediator: Pain acceptance and activity engagement (the 20-item Chronic Pain Acceptance Scale, CPAS) | Baseline (T1) to 12 weeks after post-intervention (T2) (Follow-up, T3)
  The CPAS is a validated, self-report instrument assessing pain acceptance and activity engagement. Answer format range: 0 (never true) to 6 (always true); subscale score range: 0-54 (pain acceptance subscale), 0-66 (activity engagement subscale). Higher scores yield more acceptance and activity engagement.
Mediator: Activity engagement (2 items from the 20-item Chronic Pain Acceptance Scale, CPAS) | Before each session (Ts)
  CPAS items 1 and 12 will be assessed before each session (Ts). Answer format range: 0 (never true) to 6 (always true). Higher scores yield more activity engagement.
Mediator: Activity engagement (1 item from the 20-item Chronic Pain Acceptance Scale, CPAS) | Every day for 6 days following the first session for each treatment component (Td)
  CPAS item 1 will be assessed every day for 6 days following the first session (Td) for each treatment component. Answer format range: 0 (never true) to 6 (always true). Higher scores yield more activity engagement

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zachariae, DMSc, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All data underlying publication will be shared in accordance with current data sharing regulations at host institutions.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: Researchers aiming to publish IPD meta-analyses

REFERENCES:
- [Derived] Buskbjerg C, O'Toole MS, Zachariae R, Jensen AB, Frederiksen Y, Johansen C, von Heymann A, Speckens A, Johannsen M. Optimising psychological treatment for pain after breast cancer: a factorial design study protocol in Denmark. BMJ Open. 2023 Mar 22;13(3):e066505. doi: 10.1136/bmjopen-2022-066505. PMID 36948567